CLINICAL TRIAL: NCT05025488
Title: A Phase I Open Label Peptide Based Vaccine in Patients With Myeloproliferative Neoplasm Harboring CALR Mutations
Brief Title: Mutant CALR-peptide Based Vaccine in Patients With Mutated CALR Myeloproliferative Neoplasm
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marina Kremyanskaya (Other)
Responsible Party: Sponsor-Investigator, Marina Kremyanskaya, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 22-1330
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Myelofibrosis; Essential Thrombocythemia; MPN
Keywords: CALR; Vaccine; MF; ET; peptide
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocythemia, Essential | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CALR mutated (Experimental): peptide-based vaccine in patients with myeloproliferative neoplasm (myelofibrosis and essential thrombocythemia) with CALR mutations
  Interventions: Drug: Peptide-based vaccine; Drug: Poly ICLC

INTERVENTIONS:
Drug: Peptide-based vaccine — ten (10) doses of Mutant-CALR peptides with KLH as helper peptide (in the first vaccine only). Mutant-CALR vaccine will administered every 2 weeks for the first 4 doses and then every 4 weeks for additional 6 doses. Maintenance Treatment The protocol allows for a continued administration of up to four (4) additional Mutant-CALR vaccine and four (4) Poly-ICLC administrations, 12 weeks apart.
Drug: Poly ICLC — ten (10) doses of Poly-ICLC. Poly-ICLC will be given on weeks 1, 3, 5, 7, 11, 15, 19, 23, 27 and 31. each Poly-ICLC dose must be given the day after the corresponding Mut-CALR vaccination.

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of administrating mutated-CALR peptide Vaccine to patients with MPN. The researchers plan to enroll 10 patients over a 12 month period. Maximum length of participation in 80 weeks. Patients will be asked to complete questionnaires, bone marrow biopsies, research lab collection, and standard of care lab draw. This research will be taking place only at The Mount Sinai Hospital, specifically at the Ruttenberg Treatment Center.

DETAILED DESCRIPTION:
Current MPN treatments are geared towards symptom palliation and not on changing the natural course of the disease. Mutations in calreticulin gene (CALR) is the second most common driver mutation in ET and MF patients (30%). All CALR mutations identified to date in MPN patients result in the formation of an altered protein with an identical 36-amino acid sequence in the C-terminus. This altered protein results in a MPN-specific shared neo-antigen. The mutated CALR neoantigen present in patient with MPN represents an ideal antigen for targeted immunotherapy as it is stably and specifically expressed by the malignant cells and is absent in the normal tissues. CALR neoantigen is immunogenic, effector T cells are capable of recognizing this neo-antigen, and hematopoietic cells carrying the mutation can be potently killed by these specific effector T-cells in vitro.

The researchers believe that a mutated-CALR vaccine will enhance mutated-CALR-specific T cell immunity in MPN patients carrying CALR mutations, which in turn would target and eliminate CALR+ malignant cells, thereby leading to improved clinical outcomes in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥18 years of age at the time of signing the informed consent form.
* Confirmed diagnosis of chronic phase MPN:
* Previously treated or relapsed/refectory high risk ET
* Low to intermediate 1 risk (DIPSS 0-1) PMF or ET-MF
* Verified mutation in CALR exon 9
* PS ≤ 2
* Adequate organ function:

  * Absolute neutrophil count ≥ 1000/mm3,
  * Platelet count ≥ 50,000/mm3,
  * Creatinine ≤ 2.5 mg/dL,
  * Total bilirubin ≤ 2 mg/dL, (except in patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL)
  * Transaminases < 3 times above the upper limits of the institutional normal.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to starting study medication and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks prior to first dose of vaccine. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a condom during sexual contact with a female of childbearing potential even if they have had a successful vasectomy.
* Ability to understand and the willingness to sign a written informed consent.
* Ability to adhere to the study visit schedule and all protocol requirements.
* Subjects receiving cytoreductive therapy with hydroxyurea must be on a stable dose for at least 8 weeks prior to week 1.

Exclusion Criteria:

* Other invasive malignancy in the past 3 years except non-melanoma skin cancer, localized cured prostate cancer and early stage breast cancer on HRT.
* Active autoimmune disease.
* Uncontrolled serious infection.
* Known immunodeficiency.
* Pregnant and breastfeeding women.
* Not willing to use contraception.
* Current use of immunosuppressive medications including steroids.
* Current JAK inhibitor use.
* Current use of IFN (use of anagrelide is permitted).
* Treatment with other experimental drugs within 30 days of week 1.
* Treatment with any MPN directed therapy unless otherwise noted within 5 half-lives of week 1.
* Any significant psychiatric/medical condition per investigators judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) | 32 weeks
  The Dose Limiting Toxicity (DLT) rate, defined as the proportion of patients with at least 1 grade 3 or higher AE considered to be at least possibly related to the treatment with Poly ICLC and CALR vaccines.

SECONDARY OUTCOMES:
Number of Adverse Events | Week 32
  The type, incidence, severity, seriousness, and relatedness of adverse events (AEs) per NCI CTCAE v5.0.
Number of laboratory abnormalities | Baseline through Week 32
  Number of observations, severity, and relatedness of clinical laboratory tests (hematology, biochemistry)
Change in Immune Milieu Composite | Baseline through Weeks 55 or 80
  Changes in the immune milieu (which is a composite of expression of cytokines, presence of antibodies, alterations in number and phenotype of immune cells and induction of vaccine-specific T cell response) due to the vaccines as compared to baseline values.
Change in CALR VAF | Baseline through Weeks 55 or 80
  The % change in driver mutation burden (CALR VAF) as compared to baseline
Proportion of participants who normalize their platelet number | Week 32 and weeks 55 or 80
  The proportion of patients who normalize their platelet number and/or achieve platelets less than 600 if started with platelet above 600.
Proportion of participants achieving response | Baseline and Week 32
  The proportion of patients achieving response or improvement in their disease status by ELN/IWG criteria for the categories: Complete Response; Partial Response; Clinical Improvement and Stable Disease
Myelofibrosis Symptom Assessment Form (MF-SAFv4.0) | Week 32 and weeks 55 or 80
  The proportion of patients who achieve improvement in quality of life as assessed by the by the Myelofibrosis Symptom Assessment Form. Each of the items are scored 0 to 10, with total score from 0 to 100, with higher score indicating more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Kremyanskaya, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Nina Bhardwaj, MD, PhD, Study Chair — Icahn School of Medicine at Mount Sinai; Camelia Iancu-Rubin, PhD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not determined at this time